CLINICAL TRIAL: NCT00673556
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter Study Examining the Efficacy and Safety of Weekly Intramuscular Administration of 15mg Alefacept Over 12 Weeks in a Population of Psoriasis Patients for Whom Conventional Treatment is Ineffective or Inappropriate
Brief Title: A Study to Assess the Efficacy and Safety of Alefacept in Psoriasis Patients for Whom Conventional Treatment is Ineffective or Inappropriate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-740
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Chronic Plaque Psoriasis; Alefacept
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Course A1 (Experimental)
  Interventions: Drug: alefacept
- Course A2 (Placebo Comparator)
  Interventions: Drug: placebo
- Course B (Experimental): Open label extension
  Interventions: Drug: alefacept

INTERVENTIONS:
Drug: alefacept — Intramuscular (IM)
  Other Names: Amevive; ASP0485
  Arms: Course A1; Course B
Drug: placebo — Intramuscular (IM)
  Arms: Course A2

SUMMARY:
To assess the efficacy and safety of Alefacept compared to placebo for the treatment of Chronic Plaque Psoriasis in patients for whom conventional therapies are ineffective and inappropriate

DETAILED DESCRIPTION:
Patients who completed the initial 24-week treatment course (12 weeks of weekly dosing following b y 12 weeks of follow-up) and met the eligibility criteria continued in the 24-week open label extension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Plaque Psoriasis involving ≥ 10% body surface area
* Treatment history for Psoriasis in which 3 or more conventional anti-psoriatic therapies are inappropriate or ineffective
* CD4+ T lymphocyte counts at or above the lower limit of normal

Exclusion Criteria:

* Clinically significant abnormal hematology values or blood chemistry values
* AST or ALT ≥ 3x the upper limit of normal
* Other types of Psoriasis
* Serious infection within the 3 months prior to the first dose of study drug
* History of drug or alcohol abuse within the past 2 years
* Antibody positive for HIV
* History of malignancy
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease
* Exposure to psoriasis-modifying phototherapy or high-potency topical corticosteroid therapy within 2 weeks prior to the first dose of study drug
* Exposure to systemic anti-psoriatic therapy , topical immunomodulators or topical CNIs within 4 weeks prior to the first dose of study drug
* Current treatment with any therapy for tuberculosis
* Previous exposure to Alefacept
* Nursing mothers, pregnant women, and women planning to become pregnant during the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2003-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a Psoriasis Area and Severity Index (PASI) score of ≥ 50 | 14 Weeks

SECONDARY OUTCOMES:
Proportion of patients achieving a PASI score of ≥ 50 any time during study | Throughout study
Proportion of patients achieving a PASI score of ≥ 75 | 14 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Director — Astellas Pharma US, Inc.
Locations (34):
- United States (10):
  - Irvine, California
  - Santa Monica, California
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Winston-Salem, North Carolina
  - Goodlettsville, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
- Vienna, Austria
- Belgium (3):
  - Brussels
  - Edegem
  - Liège
- Canada (9):
  - Edmonton, Alberta
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Concord, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Germany (11):
  - Bochum
  - Dresden
  - Düsseldorf
  - Essen
  - Frankfurt
  - Göttingen
  - Hamburg
  - Hanover
  - Homburg-Saar
  - Mannheim
  - Münster